CLINICAL TRIAL: NCT02646930
Title: The Impact of Chronic Endometritis on IVF Pregnancy and Pregnancy Loss Rates
Brief Title: Chronic Endometritis and IVF
Acronym: CEIVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00067725
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Chronic Endometritis; in Vitro Fertilization
Keywords: chronic endometritis; invitro fertilization; spontaneous abortion
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Incidence of CE (Experimental): To determine rates of CE in women undergoing initial IVF and outcomes
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy in women undergoing first IVF cycle

SUMMARY:
Background: Embryo quality is known to be a very important determinant to predict the implantation and pregnancy rate in IVF patients, however, the role of uterine integrity or endometrial receptivity cannot be overlooked.

Chronic endometritis (CE) is an inflammation of the endometrium diagnosed by the presence of plasma cells in the endometrial stroma. There is not only no census on the definition of CE, the current literature on the impact of CE on reproductive outcome is controversial and consists only of retrospective studies with small sample sizes. Although there is a presumption that CE is related to poor IVF outcome, this belief has not been proven.

Design: Prospective cohort study

Setting: Infertility clinics of 2 academic medical centers

Patients: Patients between the ages of ≥ 21 and ≤ 35 years old undergoing their first IVF cycle will be invited to participate.

Main Outcome Measures: The primary outcome will be ongoing pregnancy after 12 weeks estimated gestational age (EGA) with previously documented fetal cardiac motion. Secondary outcomes will include pregnancy loss rate as defined by chemical pregnancy, blighted ovum or loss of fetal cardiac motion before 12 weeks EGA.

Materials and Methods: The cycle prior to IVF, patients will undergo an in-office endometrial biopsy on cycle days 19-24. Samples will be stained for CD138 and the number of plasma cells will be quantified. The number of plasma cells in a sample that yields the best sensitivity and specificity for pregnancy will be determined by a Receiver-Operator-Curve. This number will then be used as a dichotomous variable to assign categories of "positive for CE" and "negative for CE." Pregnancy and miscarriage rates will then be determined in the positive and negative CE sample with Chi Square Analysis. A secondary sub analysis will be performed to determine pregnancy and miscarriage rates in patients who declined to participate in the study.

Expected Results: The investigators hypothesize that higher rates of CE will be found in women failing to conceive with IVF and with subsequent first-trimester miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 21 and ≤ 35 years old
* undergoing first IVF cycle
* a diagnosis of ovulatory dysfunction, pelvic factor, male factor, cervical factor or unexplained infertility

Exclusion Criteria:

* BMI > 40 kg/m2, anti-mullerian hormone (AMH) < 1.0 ng/mL or antral follicle count <10
* previous endometrial ablation
* previous uterine artery embolization
* presence of type 0, 1, 2, 3 fibroid tumor
* presence of type 4 fibroid tumor with a mean diameter of > 4 cm
* presence of uterine anomaly other than arcuate configuration
* presence of an endometrial polyp or endometrial synechiae
* presence of a hydrosalpinx on hysterosalpingography or ultrasound
* positive gonorrhea and chlamydia DNA testing
* Patients on chronic glucocorticoids (except nasal preparations), or using glucocorticoids for assisted hatching will be excluded.
* Patients on monoclonal antibody preparations directed to TNFα will be excluded.
* Post-enrollment exclusion will include patients receiving any antibiotics, except prophylaxis for transvaginal oocyte retrieval (TVOR) or glucocorticoids, except nasal preparations, from the time of endometrial biopsy until initial transvaginal ultrasound (TVUS) for pregnancy.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks gestation

SECONDARY OUTCOMES:
Implantation rate | 12 weeks
Pregnancy loss rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Price, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of Illinois, Chicago, Illinois
  - Duke Fertility Clinic, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided